CLINICAL TRIAL: NCT04757363
Title: A Phase II Study of Nivolumab in Combination With FOLFOX and Regorafenib in Patients With HER2-Negative Metastatic Esophagogastric Cancer
Brief Title: A Study of Nivolumab Combined With FOLFOX and Regorafenib in People Who Have HER2-Negative Esophagogastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-540
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Esophagogastric Cancer; HER2-Negative
Keywords: nivolumab (OPDIVO®); regorafenib (STIVARGA®); fluorouracil; leucovorin; oxaliplatin; Regorafenib; esophageal cancer; 20-540
MeSH Terms: conditions — Esophageal Neoplasms | interventions — regorafenib; Nivolumab; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, nonrandomized, single-institution, phase II study of nivolumab in combination with FOLFOX and regorafenib as first-line therapy in patients with metastatic esophagogastric adenocarcinoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab Combined With FOLFOX and Regorafenib (Experimental): Each treatment cycle consists of 28 days. Patients will initially receive induction therapy with regorafenib (80 mg on days 1-21 of the 28-day cycle) and nivolumab (240 mg on days 1 and 15 of the 28-day cycle). Starting on cycle 2, day 1, patients will also receive FOLFOX chemotherapy with oxaliplatin (85 mg/m2 IV), leucovorin (400 mg/m2 IV), 5-FU (400 mg/m2 IV bolus), and 5-FU (2400 mg/m2/day continuous IV infusion over 48 h). If the patient is not a good candidate for induction regorafenib and nivolumab (i.e. symptomatic from a large burden of disease), 5-FU and oxaliplatin can be added during cycle 1 at the treating physician's discretion. 39 Patients will continue with this regimen until disease progression, unacceptable toxicity, or development of serious intercurrent illness. Treatment will be performed on the scheduled day (±7-day treatment window).
  Interventions: Drug: regorafenib; Drug: nivolumab; Drug: FOLFOX chemotherapy with oxaliplatin

INTERVENTIONS:
Drug: regorafenib — regorafenib (80 mg on days 1-21 of the 28-day cycle)
Drug: nivolumab — nivolumab (240 mg on days 1 and 15 of the 28-day cycle).
Drug: FOLFOX chemotherapy with oxaliplatin — FOLFOX chemotherapy with oxaliplatin (85 mg/m2 IV), leucovorin (400 mg/m2 IV), 5-FU (400 mg/m2 IV bolus), and 5-FU (2400 mg/m2/day continuous IV infusion over 48 h).

SUMMARY:
The purpose of this study is to find out whether combining nivolumab, FOLFOX, and regorafenib may be a safe and effective treatment for people who have HER2-negative metastatic esophagogastric cancer.

Nivolumab is an antibody, like the proteins made by the immune system to protect the body from harm. Nivolumab blocks the protein PD-1 (programmed cell death receptor-1) that usually acts as a "brake" on the immune system. Blocking this protein is like releasing the brakes, so that the immune system can target cancer cells and destroy them.

FOLFOX is a combination of three standard chemotherapy drugs (leucovorin, 5-fluorouracil, and oxaliplatin) commonly used to treat your type of cancer. The drugs work by damaging the DNA in cancer cells, which can cause the cells to stop growing and die.

Regorafenib is a type of drug called a tyrosine kinase inhibitor (TKI). This drug targets the tyrosine kinase protein found in or on the surface of cancer cells that the cells need to survive and grow. Blocking this protein may stop cancer cells from growing, or cause them to grow more slowly or to shrink.

The study researchers think that combining nivolumab, FOLFOX, and regorafenib may be a more effective treatment for HER2-negative metastatic esophagogastric cancer than the usual chemotherapy treatment(s) alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic esophageal, gastric, or gastroesophageal junction adenocarcinoma
* Patients must have disease that can be evaluated radiographically within 28 days of the start of study treatment. This may be measurable disease or non-measurable disease per RECIST 1.1.
* Age 18 years or older
* ECOG performance status 0 to 1
* Peripheral neuropathy grade ≤1
* Available archival tissue for correlative analysis (biopsy is required if no archival tissue is available)
* Adequate organ function as below:

  * Absolute neutrophil count ≥1500/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥9 g/dL
  * Serum creatinine ≤1.5X ULN
  * Serum total bilirubin ≤1.5X ULN OR Direct bilirubin ≤ULN for s ubjects with total bilirubin levels >1.5X ULN, except patients with Gilbert's disease (≤3X ULN)
  * AST and ALT ≤2.5X ULN
  * Albumin ≥3 mg/dL
  * ALT, alanine aminotransferase; AST, aminotransferase; ULN, upper limit of normal.

Exclusion Criteria:

* Confirmed HER2-positive disease (IHC 3+ or 2+, fluorescence in situ hybridization HER2:CEP17 ratio ≥2)

  ° Note: Participants that are IHC 2+ but negative by FSH w ill be considered HER2- negative and eligible for trial.
* Inability to swallow oral pills
* Prior chemotherapy for metastatic disease. Patients with metastatic disease after treatment for localized esophagogastric cancer may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if >6 months have elapsed between the end of adjuvant therapy and registration
* Currently participating in a study and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Underwent major surgical procedure within 4 weeks of registration
* Underwent radiation within 2 weeks of registration
* Received prior therapy with regorafenib
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Diagnosis of immunodeficiency or receipt of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of trial treatment
* A known history of active Bacillus tuberculosis
* A known active central nervous system metastases and/or carcinomatous meningitis
* A known history of or any evidence of active, noninfectious pneumonitis
* An active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, systemic lupus erythematosus, Wegener syndrome [granulomatosis with polyangiitis], myasthenia gravis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis) within the 3 years before the start of treatment. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
* A known history of human immunodeficiency virus (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients with HBsAg reactive on entecavir may be eligible after consultation with hepatologist and study team.
* Received a live vaccine within 30 days of planned start of study therapy
* Active or clinically significant cardiac disease, including congestive heart failure-New York Heart Association class >II, active coronary artery disease, cardiac arrhythmias requiring antiarrhythmic therapy other than beta blockers or digoxin, unstable angina (anginal symptoms at rest), new-onset angina within 3 months before initiation, or myocardial infarction within 6 months before initiation
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure >90 mm Hg on repeated measurement) despite optimal medical management
* Evidence or history of bleeding diathesis or coagulopathy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment
* Unwilling to give written, informed consent, unwilling to participate, or unable to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
6-month progression free Survival | 6 months
  will be defined according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Cytryn SL, Moy RH, Cowzer D, Shah RH, Chou JF, Joshi SS, Ku GY, Maron SB, Desai A, Yang J, Sugarman R, Rao D, Goldberg Z, Charalambous C, Lapshina M, Antoine A, Socolow F, Trivedi N, Capanu M, Gerdes H, Schattner MA, Simmons M, Lacouture ME, Paroder V, Tang LH, Shia J, Ilson DH, Solit DB, Berger MF, Janjigian YY. First-line regorafenib with nivolumab and chemotherapy in advanced oesophageal, gastric, or gastro-oesophageal junction cancer in the USA: a single-arm, single-centre, phase 2 trial. Lancet Oncol. 2023 Oct;24(10):1073-1082. doi: 10.1016/S1470-2045(23)00358-3. Epub 2023 Sep 1. PMID 37666264
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm